CLINICAL TRIAL: NCT05242614
Title: The Effects of a Hybrid Face-To-Face and Online Mode of Delivering a Mindfulness-Based Dementia Caregiving Programme for Family Caregivers of Persons With Dementia: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Dr. Kor Pui Kin Patrick, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20210709005
Record Dates: First submitted 2022-02-08; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This study is a two-arm parallel randomized controlled trial, with an intervention group (mindfulness group) and a control group. The participants in the MBI group will receive 6 weekly 90-minute group-based sessions delivered through a face-to-face and online approach. The participants in control group will receive brief education on dementia care with the same group size, duration, and frequency as the sessions in the intervention group.
Who Masked: Outcomes Assessor
Masking Description: All outcome measurements will be collected by an independent trained assessor (a trained research assistant) who are blinded to the group assignment of the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A hybrid Mindfulness-based Dementia Caregiving Program (MBDCP) (Experimental): Participants from the experimental group will receive a hybrid Mindfulness-based Dementia Caregiving Program (MBDCP). It is a 6-week program. In the 1st, 2nd and 6th session, it is delivered through face to face, while in the 3rd, 4th and 5th sessions, it will be delivered via online approach.
  Interventions: Behavioral: The Hybrid Mindfulness-based Dementia caregiving program (MBDCP)
- Control group (Active Comparator): The family caregivers in the control group will receive 6 week education programme on dementia. It is a control for the social effects of the MBDCP. In the 1st, 2nd and 6th session, it is delivered through face to face, while in the 3rd, 4th and 5th sessions, it will be delivered via online approach.
  Interventions: Behavioral: Psychoeducation educational program

INTERVENTIONS:
Behavioral: The Hybrid Mindfulness-based Dementia caregiving program (MBDCP) — The hybrid MBDCP includes 6 weekly 90-minute group-based sessions delivered through a face-to-face (1st, 2nd, and 6th sessions) and online approach (3rd, 4th, and 5th sessions). The online session is designed for self-directed learning. The MBDCP includes different mindfulness practices (e.g., mindful eating, body scanning, and mindful walking), psychoeducation on caregiving, and group sharing, aimed at helping caregivers to develop mindfulness skills through the formal and informal practice of mindfulness, and to integrate these skills into their everyday life. The duration of each session is 90 minutes. Th MBDCP will be delivered by a qualified mindfulness therapist. In the MBDCP's online sessions, the caregivers will watch a teaching video (e.g., a video demonstrating mindfulness practices) through a website.
  Arms: A hybrid Mindfulness-based Dementia Caregiving Program (MBDCP)
Behavioral: Psychoeducation educational program — This program serves as a control for the social effects of the MBDCP. The brief education program consists of 6 weekly 90-minutes group sessions in which the sessions (1st, 2nd, and 6th) and (3rd 4th 5th) will be delivered through the face-to-face and online approach respectively, with the similar group size of the MBDCP. The education contents include caregiving skills, education on mood, and group sharing. The program will be led by a nurse.
  Arms: Control group

SUMMARY:
Mindfulness-based intervention (MBI) has been shown promising effects in enhancing the well-being of caregivers of patients with dementia (PWD). However, the time schedule and the mode of delivering the conventional MBI was demanding to family caregivers of PWD, and therefore impeding the feasibility of use among caregivers. Our research team had developed a hybrid MBI program which includes face to face and online mode of mindfulness sessions w. The study aims to evaluate the effectiveness of this 6-week hybrid MBI program on caregivers of PWD over a 6-month follow up. This study is a two-arm parallel randomized controlled trial. Participants are family caregivers of PWD and we aimed to recruit 290 subjects. Eligible participants will be recruited from three local nongovernmental organizations (NGOs) in Hong Kong. They will be randomly allocated into MBI group and a control group (with 145 participants in each group) . The participants in the MBI group will receive 6 weekly 90-minute group-based sessions delivered through a face-to-face and online approach. The participants in control group will receive brief education on dementia care with the same group size, duration, and frequency as the sessions in the intervention group. Assessment (using questionnaire) about caregiving stress and other outcomes (positive aspect of caregiving, depression, dyadic relationship, anxiety, neuropsychiatric symptoms of patients) will be assessed at baseline, immediately after the intervention and at the 6-month follow up. Focus group interview will also be conducted to explore family caregivers' experience in participating in the program. We aimed to recruit 20 caregivers for the interviews via purposive sampling. It is hypothesized that compared to the control group, the MBI group will have a reduction on caregiving stress and improve other outcomes after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers who are aged 18 or above
* Caregivers who are taking care for a family member medically diagnosed with dementia who has been residing in the community;
* Caregivers who are providing care to the dementia care recipients for at least 6 months prior to the subject recruitment.

Exclusion Criteria:

* Caregivers who have participated in any structured psychosocial intervention or mindfulness-based intervention/training in the 6 months prior to recruitment,
* Caregivers who have acute psychiatric and medical comorbidities that are potentially life-threatening (e.g., suicidal ideation) or leave them with a limited ability to participate or adhere to the intervention (e.g., acute psychosis),
* caregivers who do not have Internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in perceived Stress scale of caregivers | baseline, immediately after the intervention, 6 month- after the intervention
  The change in stress will be measured by the Chinese version of perceived stress scale (Cohen et al., 1983) . The PSS contains 10 items. It is a 5 point Likert scale (1= never, 5=Very often). The total score is ranged from 10 to 50. A higher score indicating higher level of perceived stress

SECONDARY OUTCOMES:
Change in depressive symptoms of caregivers | baseline, immediately after the intervention, 6 month- after the intervention
  The change in depressive symptoms will be measured by the Centre for Epidemiologic Studies Depression scale (CESD) (Robert & Vernon, 1983) . It is a self-reported measurement containing 20 items. Rating were based on a 4 point likert scale ranging from 0 (Rarely or none of the time) to 3 (most or all of the time). The total score is ranged from 0-60. A higher score indicates a higher level of depression
Change in positive caregiving experience of caregivers | baseline, immediately after the intervention, 6 month- after the intervention
  This will be measured by thePositive aspect of caregiving scale (PAC) (Kate et al., 2012) . The PAC contains 11 items with 5 point likert scale for all item responses. The total score ranged from 11 to 55. , with higher score indicating a more positive perception of caregiving.
Change in caregiving burden of caregivers | baseline, immediately after the intervention, 6 month- after the intervention
  This will be measured by the Zarit Burden Interview (ZBI) (Zarit et al,1980) . The scale comprises of 22 items. Items are presented in the format of 5 point Likert scale (0= None, 4=Extremely distressing). The total score is ranged from 0-88, with a higher score representing a higher level of caregiving burden.
Change in dyadic relationship | baseline, immediately after the intervention, 6 month- after the intervention
  This will be measured using the dyadic relationship scale(Sebern & Whitlatch, 2007). This scale is completed by the family caregivers and it assesses a variety of relationship stressor. Items are presented in a format of 4 point Likert scale (1= strongly disagree, 4 =strongly agree). The scale contains two subscale scores: dyadic strain (range of score: 5-20) and positive dyadic relationship (range of score: 6 to 24) . Higher score on each of these scales indicate higher level of strain and positive interactions respectively.
Change in heart rate variability of caregivers | baseline, immediately after the intervention, 6 month- after the intervention
  This will be measured by using validated Polar heart rate monitors. Heart rate variability will be interpreted following the guidelines for the Standard measurement and interpretation of HRV (European Society of Cardiology and the North American Society of Pacing and Electrophysiology) using the frequency domain method ( Vanderlei et al 2008; Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology, 1996).
Change in neuropsychiatric symptoms of the care recipients | baseline, immediately after the intervention, 6 month- after the intervention
  This will be measured by the Neuropsychiatric inventory Questionnaire (NPI-Q) (Cummings et al., 1994) through caregivers. NPI-Q is an informant based instrument that measures the presence and severity of 12 symptoms in patients with dementia and caregivers distress. The caregivers will be asked to identify whether the symptoms of the care recipients had been present in the past week, and rate the severity of the symptoms (from a likert scale ranged from 1 to 3) and the corresponding distress to them( from likert scale ranged from 1 to 5). The NPI-Q provides two scores, namely, total severity of symptoms (range of score: 12 to 36) and total distress scores (range of score: 12 to 60). The higher scores of these two subscales represent a higher level of symptoms severity of care recipients and distress of caregivers.

OTHER OUTCOMES:
Level of mindfulness | baseline, immediately after the intervention, 6 month- after the intervention
  Caregivers' level of mindfulness will be measured as the process indicator by using the Five Facets Mindfulness Questionnaire Short Form (Baer et al., 2006) . It is a 20 item self-report questionnaire measuring the five facets of mindfulness which includes observing, describing, acting with awareness, non-judging of inner and non-reactivity to inner experience. The total score ranges from 20 to 100 and the higher the score, the higher level of mindfulness.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Roberts RE, Vernon SW. The Center for Epidemiologic Studies Depression Scale: its use in a community sample. Am J Psychiatry. 1983 Jan;140(1):41-6. doi: 10.1176/ajp.140.1.41. PMID 6847983
- [Background] Kate N, Grover S, Kulhara P, Nehra R. Scale for positive aspects of caregiving experience: development, reliability, and factor structure. East Asian Arch Psychiatry. 2012 Jun;22(2):62-9. PMID 22714876
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628
- [Background] Vanderlei LC, Silva RA, Pastre CM, Azevedo FM, Godoy MF. Comparison of the Polar S810i monitor and the ECG for the analysis of heart rate variability in the time and frequency domains. Braz J Med Biol Res. 2008 Oct;41(10):854-9. doi: 10.1590/s0100-879x2008005000039. Epub 2008 Sep 30. PMID 18853042
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Derived] Kor PPK, Li ML, Kwok DKS, Leung AYM, Lai DLL, Liu JYW. Evaluating the effectiveness of a 6-week hybrid mindfulness-based intervention in reducing the stress among caregivers of patients with dementia during COVID-19 pandemic: protocol of a randomized controlled trial. BMC Psychol. 2022 Jul 19;10(1):178. doi: 10.1186/s40359-022-00876-8. PMID 35854347